CLINICAL TRIAL: NCT07105683
Title: Effect of Kinetic Control Training on Postnatal Low Back Pain
Acronym: KCT-PLBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Ahmed Mohammed, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005122; P.T.REC/012/005122 (Other: Ethical committe faculty of physical therapy CU)
Record Dates: First submitted 2025-07-04; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot Pack Therapy Only (Control Group) (Active Comparator): Participants in this arm receive hot pack therapy as a standard physiotherapeutic intervention. A moist hot pack is applied to the lumbar region for 20-30minutes per session, twice daily, over a period of 8weeks. This intervention is intended to provide superficial heat to reduce pain, promote muscle relaxation, and improve local circulation. No additional therapeutic exercises are administered to this group
  Interventions: Other: hot pack therapy
- Hot Pack Therapy + Kinetic Control Training (Experimental Group) (Experimental): Participants in this arm receive both hot pack therapy and kinetic control training. The hot pack is applied to the lumbar region for 20-30minutes per session, twice daily, for 8weeks. In addition, participants undergo kinetic control training, which includes therapist-guided exercises targeting the deep stabilizing muscles of the lumbar-pelvic region. Exercises focus on improving muscle coordination, movement control, and spinal stability. Sessions are conducted three times per week for 8 weeks.
  Interventions: Other: hot pack therapy; Genetic: Kinetic control training

INTERVENTIONS:
Other: hot pack therapy — Application of a commercial hot pack to the lumbar region for 20-30 minutes per session, twice daily, for 6 weeks.
Genetic: Kinetic control training — is an evidence-based rehabilitation approach, focused on retraining movement patterns by addressing and improving motor control of the lumbar spine and pelvis, correcting faulty movement strategies, enhancing stability in functional tasks. The principles of KCT entail the identification of direction-specific motor control deficit, uncontrolled extension, followed by focused retraining of movement control through specific exercises designed to improve the coordination and activation of deep stabilizing muscle systems, including the transversus abdominis, multifidus, and pelvic floor muscles. This approach is especially relevant in postpartum women, where motor control deficits and poor load transfer capabilities are commonly observed . Based on the clinical presentation of patients with postnatal low back pain, demonstrated symptoms that were aggravated during lumbar extension movements or when maintaining prolonged upright postures. The
  Arms: Hot Pack Therapy + Kinetic Control Training (Experimental Group)

SUMMARY:
the effect of kinetic control training and hotpack and compare it with hotpack alone on postnatal low back pain

DETAILED DESCRIPTION:
Background: Postnatal low back pain (PLBP) is a common condition affecting women after childbirth due to musculoskeletal and biomechanical changes during pregnancy. Effective rehabilitation strategies are essential for pain relief and functional recovery.

Objective: This study aims to evaluate the effect of kinetic control training in postnatal women with low back pain.

Methods: A total of 66 postnatal women with low back pain were randomly selected from WENGAT Hospital and EL SHATBY Hospital in Alexandria. Participants were divided into two equal groups:

Group A: 33 women treated with hot pack for 20 minutes twice daily for 6 weeks. Group B: 33 women treated with a combination of kinetic control training and hot pack 3 sessions/week for 6 weeks.

Pain intensity will be assessed using the Visual Analog Scale (VAS) and Pressure Algometer. Range of motion (ROM) will be evaluated using the Modified Schober Test.

ELIGIBILITY:
**Inclusion Criteria:**

* Female patients with postnatal low back pain (PLBP) that lasted for at least 6 months.
* Pain intensity ≥ 5 on the Visual Analog Scale (VAS).
* Limitation score ≤ 5 on the Modified Schober Test.
* Age between 25 and 35 years.
* Body mass index (BMI) between 20-25 kg/m².
* Medically stable and able to provide informed consent.
* Positive result in the extension uncontrolled movement test, indicating:
* Loss of lumbopelvic control.
* Overactivity of global extensors during functional tasks. *Exclusion Criteria:**
* Any neurological or rheumatological disorders.
* Previous spinal surgery.
* Pregnancy or planning to become pregnant during the study period.
* BMI outside the 20-25 kg/m² range.
* Inability to participate in exercise or physical activity.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — **Inclusion Criteria:**
  * Female patients with postnatal low back pain (PLBP) that lasted for at least 6 months.
  * Pain intensity ≥ 5 on the Visual Analog Scale (VAS).
  * Limitation score ≤ 5 on the Modified Schober Test.
  * Age between 25 and 35 years.
  * Body mass index (BMI) between 20-25 kg/m².
  * Medically stable and able to provide informed consent.
  * Positive result in the extension uncontrolled movement test, indicating:
  * Loss of lumbopelvic control.
  * Overactivity of global extensors during functional tasks.
  **Exclusion Criteria:**
  * Any neurological or rheumatological disorders.
  * Previous spinal surgery.
  * Pregnancy or planning to become pregnant during the study period.
  * BMI outside the 20-25 kg/m² range.
  * Inability to participate in exercise or physical activity.
Enrollment: 66 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Measured by Visual Analog Scale (VAS) | Baseline and after 8weeks of intervention
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a validated tool for measuring subjective pain levels. Participants will indicate their pain level on a 10 cm horizontal line ranging from "no pain" (0) to "worst imaginable pain" (10). This measurement will help evaluate the effectiveness of kinetic control training in reducing postnatal low back pain compared to hot pack therapy alone

SECONDARY OUTCOMES:
Lumbar Range of Motion (Flexion and Extension) Using Modified Schober Test | Baseline and after 8weeks of intervention
  This measure assesses the flexibility and mobility of the lumbar spine using the Modified Schober Test. A non-invasive tape measure method is used to evaluate the difference in spinal segment length during full flexion and extension compared to the neutral standing posture. The outcome reflects the degree of lumbar mobility, which may be affected by postnatal low back pain and improved through targeted interventions like kinetic control training.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Fawzy, Phd, Principal Investigator — Om el masryen hospital
Locations (1):
- physical therapy cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The plan for sharing deidentified individual participant data is under consideration. It will depend on institutional policies and ethical approvals. Further details will be provided once finalized.

REFERENCES:
- See also: Official study information page hosted by Cairo University. — https://www.cu.edu.eg